CLINICAL TRIAL: NCT06046261
Title: Exploring the Impact of " ACP Board Game for Life" on Death Preparation and Anxiety in Patients With Stage 4 and 5 Chronic Kidney Diseases: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: B-ER-110-472
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Chronic Kidney Disease; Chronic Renal Failure; Chronic Renal Insufficiency; End of Life Care; Advance Care Planning; Death Anxiety
Keywords: Chronic Kidney Disease; Death Preparation; Death Anxiety; Advance Care Planning; Board Game
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic; Necrophobia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General routine care and ACP board game for life (Experimental)
  Interventions: Other: ACP board game for life
- General routine care (No Intervention): "General routine care" means that when a CKD stage 4-5 patient is in critical condition or at the end of life, the renal medical team will explain the content of DNR to the patient's family (without cardiopulmonary resuscitation: including endotracheal tube intubation, extracorporeal cardiac compression, Emergency treatment items such as cardiac electric shock, emergency drug injection, and artificial cardiac pacemaker adjustment), the concept of palliative care (supportive care for end-of-life patients to relieve physical discomfort symptoms to reduce physical, mental and spiritual pain) or ACP.

INTERVENTIONS:
Other: ACP board game for life — The research subjects will be assigned to the experimental group or the control group according to their wishes. Those who are willing to participate the ACP board game will be assigned to the experimental group. The intervention time for each board game is around 2 hours. There are 60 cards in this ACP board game; the focus of the game is to know the participants' thoughts on the card options. Questionnaires need to be filled in before and after intervention.
  Arms: General routine care and ACP board game for life

SUMMARY:
This study was to explore the impacts of participating in "ACP board game for life" on death preparation, death anxiety, end-of-life care preferences, and intervention perception in stage 4-5 CKD patients with advanced chronic kidney diseases in a medical center.

DETAILED DESCRIPTION:
This study was to explore the impacts of participating in "ACP board game for life" on death preparation, death anxiety, end-of-life care preferences, and intervention perception in stage 4-5 CKD patients with advanced chronic kidney diseases in a medical center. A nonrandomized two-arm pretest and posttest quasi-experimental design was used. Patients in the control group received routine care while patients in the experimental group received routine care and ACP board game for life. The ACP board game, death preparation subscale, Chinese Likert death anxiety scale, self-created questionnaires and brief interview were used for data collection.

ELIGIBILITY:
Inclusion Criteria:

* Stage 4-5 chronic kidney disease patients
* Chinese nationality
* Over 20 years old
* Consciousness clear, can communicate and express their opinions in Mandarin and Taiwanese

Exclusion Criteria:

* Patients express that talking about death makes them feel scared or cause anxiety
* The doctor assesses that the patient's condition is in the stage of septic shock, hemodynamic instability, asthma, pulmonary edema, hypoxemia or acute myocardial infarction
* Patients with contact or airborne precautions
* Patients without legal capacity

Ages: 21 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Death Preparation | 2hours
  The death preparation subscale total of 8 items measure death preparation.The range of total scores of the subscale is 8-40. It shows that the higher scores, the better death preparedness.
Death Anxiety | 2hours
  The Chinese Likert death anxiety scale was used, with a total of 15 items, using a Likert scale of 1 to 5 (1 means completely disagree, 2 means disagree, 3 means fair, 4 means agree, and 5 means completely agree) ), the total scores of the scale ranges from 15 to 75. The higher total scores, the higher degree of death anxiety.
End-of-Life Care Preferences | 2hours
  A self-made questionnaire on end-of-life care preferences for patients with stage 4-5 CKD was used. There were 2 items in the scale. The item type was multiple choice, the scoring method is based on the number of times and percentages chosen by the participants.
Intervention Perception | 2hours
  A self-made questionnaire on the feelings of CKD stage 4-5 patients after participating in the " ACP board game for life " was used. There are 4 items in the scale, using a Likert scoring method of 1 to 5 points (1 point means completely disagree, 2 points means disagree, 3 points means neither agree nor disagree, 4 points means agree, 5 points means strongly agree), the scoring method is based on the participant's options for Mean±SD, frequency and percentage statistics.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdel-Khalek AM, El Nayal MA. Death anxiety in Lebanese college students in 1998 and 2015. Death Stud. 2019;43(9):542-546. doi: 10.1080/07481187.2018.1500006. Epub 2018 Sep 5. PMID 30183514
- [Background] An E, Lo C, Hales S, Zimmermann C, Rodin G. Demoralization and death anxiety in advanced cancer. Psychooncology. 2018 Nov;27(11):2566-2572. doi: 10.1002/pon.4843. Epub 2018 Aug 20. PMID 30053317
- [Background] Ang YG, Heng BH, Saxena N, Liew STA, Chong PN. Annual all-cause mortality rate for patients with diabetic kidney disease in Singapore. J Clin Transl Endocrinol. 2016 Jan 27;4:1-6. doi: 10.1016/j.jcte.2016.01.002. eCollection 2016 Jun. PMID 29159125
- [Background] Axelsson L, Alvariza A, Lindberg J, Ohlen J, Hakanson C, Reimertz H, Furst CJ, Arestedt K. Unmet Palliative Care Needs Among Patients With End-Stage Kidney Disease: A National Registry Study About the Last Week of Life. J Pain Symptom Manage. 2018 Feb;55(2):236-244. doi: 10.1016/j.jpainsymman.2017.09.015. Epub 2017 Sep 21. PMID 28941964
- [Background] Bekker YAC, Suntjens AF, Engels Y, Schers H, Westert GP, Groenewoud AS. Advance care planning in primary care: a retrospective medical record study among patients with different illness trajectories. BMC Palliat Care. 2022 Feb 14;21(1):21. doi: 10.1186/s12904-022-00907-6. PMID 35152892
- [Background] Caserta M, Utz R, Lund D, Supiano K, Donaldson G. Cancer Caregivers' Preparedness for Loss and Bereavement Outcomes: Do Preloss Caregiver Attributes Matter? Omega (Westport). 2019 Dec;80(2):224-244. doi: 10.1177/0030222817729610. Epub 2017 Sep 8. PMID 28886674
- [Background] Chan HL, Li IF, Tseng LC, Hsiung Y. Exploring Behavioral Readiness and Program Strategies to Engage Older Community Residents in Advance Care Planning: A Pilot Mixed-Method Study in Taiwan. Int J Environ Res Public Health. 2020 Jun 16;17(12):4285. doi: 10.3390/ijerph17124285. PMID 32560049
- [Background] Chan TH, Chan FM, Tin AF, Chow AY, Chan CL. Death preparation and anxiety: a survey in Hong Kong. Omega (Westport). 2006-2007;54(1):67-78. doi: 10.2190/6478-6572-v704-1545. PMID 17844773
- [Background] Cross SH, Lakin JR, Mendu M, Mandel EI, Warraich HJ. Trends in Place of Death for Individuals With Deaths Attributed to Advanced Chronic or End-Stage Kidney Disease in the United States. J Pain Symptom Manage. 2021 Jan;61(1):112-120.e1. doi: 10.1016/j.jpainsymman.2020.08.001. Epub 2020 Aug 10. PMID 32791183
- [Background] Davison SN. End-of-life care preferences and needs: perceptions of patients with chronic kidney disease. Clin J Am Soc Nephrol. 2010 Feb;5(2):195-204. doi: 10.2215/CJN.05960809. Epub 2010 Jan 14. PMID 20089488
- [Background] Delanaye P, Jager KJ, Bokenkamp A, Christensson A, Dubourg L, Eriksen BO, Gaillard F, Gambaro G, van der Giet M, Glassock RJ, Indridason OS, van Londen M, Mariat C, Melsom T, Moranne O, Nordin G, Palsson R, Pottel H, Rule AD, Schaeffner E, Taal MW, White C, Grubb A, van den Brand JAJG. CKD: A Call for an Age-Adapted Definition. J Am Soc Nephrol. 2019 Oct;30(10):1785-1805. doi: 10.1681/ASN.2019030238. Epub 2019 Sep 10. PMID 31506289
- [Background] Deodhar J, Nagaraju SP, Kirpalani AL, Nayak AM. Shared Decision-Making, Advance Care Planning for Chronic Kidney Disease Patients. Indian J Palliat Care. 2021 May;27(Suppl 1):S33-S36. doi: 10.4103/ijpc.ijpc_71_21. Epub 2021 May 30. PMID 34188376
- [Background] Desta BZ, Dadi AF, Derseh BT. Mortality in hemodialysis patients in Ethiopia: a retrospective follow-up study in three centers. BMC Nephrol. 2023 Jan 4;24(1):3. doi: 10.1186/s12882-022-03053-6. PMID 36600194
- [Background] Douglas CA. Palliative care for patients with advance chronic kidney disease. J R Coll Physicians Edinb. 2014;44(3):224-31. doi: 10.4997/JRCPE.2014.309. PMID 25318401
- [Background] Durepos P, Sussman T, Ploeg J, Akhtar-Danesh N, Punia H, Kaasalainen S. What Does Death Preparedness Mean for Family Caregivers of Persons With Dementia? Am J Hosp Palliat Care. 2019 May;36(5):436-446. doi: 10.1177/1049909118814240. Epub 2018 Dec 5. PMID 30518228
- [Background] Galiana L, Oliver A, De Simone G, Linzitto JP, Benito E, Sanso N. A Brief Measure for the Assessment of Competence in Coping With Death: The Coping With Death Scale Short Version. J Pain Symptom Manage. 2019 Feb;57(2):209-215. doi: 10.1016/j.jpainsymman.2018.11.003. Epub 2018 Nov 15. PMID 30447381
- [Background] Gonzalez AM, Gutman T, Lopez-Vargas P, Anumudu S, Arce CM, Craig JC, Dunn L, Eckardt KU, Harris T, Levey AS, Lightstone L, Scholes-Robertson N, Shen JI, Teixeira-Pinto A, Wheeler DC, White D, Wilkie M, Jadoul M, Winkelmayer WC, Tong A. Patient and Caregiver Priorities for Outcomes in CKD: A Multinational Nominal Group Technique Study. Am J Kidney Dis. 2020 Nov;76(5):679-689. doi: 10.1053/j.ajkd.2020.03.022. Epub 2020 May 31. PMID 32492463
- [Background] Gotze H, Brahler E, Gansera L, Schnabel A, Gottschalk-Fleischer A, Kohler N. Anxiety, depression and quality of life in family caregivers of palliative cancer patients during home care and after the patient's death. Eur J Cancer Care (Engl). 2018 Mar;27(2):e12606. doi: 10.1111/ecc.12606. Epub 2016 Nov 17. PMID 27859889
- [Background] Holley JL. Palliative care in end-stage renal disease: focus on advance care planning, hospice referral, and bereavement. Semin Dial. 2005 Mar-Apr;18(2):154-6. doi: 10.1111/j.1525-139X.2005.18208.x. PMID 15771661
- [Background] Holley JL. Advance care planning in CKD/ESRD: an evolving process. Clin J Am Soc Nephrol. 2012 Jun;7(6):1033-8. doi: 10.2215/CJN.00580112. Epub 2012 Mar 29. PMID 22461536
- [Background] Holley JL, Davison SN. Advance care planning for patients with advanced CKD: a need to move forward. Clin J Am Soc Nephrol. 2015 Mar 6;10(3):344-6. doi: 10.2215/CJN.00290115. Epub 2015 Feb 13. No abstract available. PMID 25680738
- [Background] Hong YA, Chung S, Park WY, Bae EJ, Yang JW, Shin DH, Kim SW, Shin SJ; Committee on Ethical Issues of the Korean Society of Nephrology. Nephrologists' Perspectives on Decision Making About Life-Sustaining Treatment and Palliative Care at End of Life: A Questionnaire Survey in Korea. J Palliat Med. 2021 Apr;24(4):527-535. doi: 10.1089/jpm.2020.0248. Epub 2020 Sep 30. PMID 32996855
- [Background] Hovland C. When Death With Dementia Is "A Memory Seared in My Brain": Caregivers' Recommendations to Health Care Professionals. J Appl Gerontol. 2020 Nov;39(11):1195-1202. doi: 10.1177/0733464819884267. Epub 2019 Oct 23. PMID 31640462
- [Background] Hovland CA, Kramer BJ. Barriers and Facilitators to Preparedness for Death: Experiences of Family Caregivers of Elders with Dementia. J Soc Work End Life Palliat Care. 2019 Jan-Mar;15(1):55-74. doi: 10.1080/15524256.2019.1595811. Epub 2019 Apr 18. PMID 30995886
- [Background] Khodarahimi S, Veiskarami HA, Mazraeh N, Sheikhi S, Rahimian Bougar M. Mental Health, Social Support, and Death Anxiety in Patients With Chronic Kidney Failure. J Nerv Ment Dis. 2021 Nov 1;209(11):809-813. doi: 10.1097/NMD.0000000000001386. PMID 34238892
- [Background] Ladin K, Neckermann I, D'Arcangelo N, Koch-Weser S, Wong JB, Gordon EJ, Rossi A, Rifkin D, Isakova T, Weiner DE. Advance Care Planning in Older Adults with CKD: Patient, Care Partner, and Clinician Perspectives. J Am Soc Nephrol. 2021 Jun 1;32(6):1527-1535. doi: 10.1681/ASN.2020091298. Epub 2021 Apr 7. PMID 33827902
- [Background] Liu L, Chan HY, Ho TC, Chow RS, Li MM, Cheung EW, Gu C, Wang Y. A serious game for engaging older adults in end-of-life care discussion: A mixed method study. Patient Educ Couns. 2023 Aug;113:107787. doi: 10.1016/j.pec.2023.107787. Epub 2023 May 3. PMID 37148841
- [Background] Liu L, Zhao YY, Yang C, Chan HY. Gamification for promoting advance care planning: A mixed-method systematic review and meta-analysis. Palliat Med. 2021 Jun;35(6):1005-1019. doi: 10.1177/02692163211005343. Epub 2021 Mar 29. PMID 33775174
- [Background] Loosman WL, Rottier MA, Honig A, Siegert CE. Association of depressive and anxiety symptoms with adverse events in Dutch chronic kidney disease patients: a prospective cohort study. BMC Nephrol. 2015 Sep 21;16:155. doi: 10.1186/s12882-015-0149-7. PMID 26390864
- [Background] Luckett T, Spencer L, Morton RL, Pollock CA, Lam L, Silvester W, Sellars M, Detering KM, Butow PN, Tong A, Clayton JM. Advance care planning in chronic kidney disease: A survey of current practice in Australia. Nephrology (Carlton). 2017 Feb;22(2):139-149. doi: 10.1111/nep.12743. PMID 26860214
- [Background] Maddalena V, O'Shea F, Barrett B. An Exploration of Palliative Care Needs of People With End-Stage Renal Disease on Dialysis: Family Caregiver's Perspectives. J Palliat Care. 2018 Jan;33(1):19-25. doi: 10.1177/0825859717747340. Epub 2017 Dec 27. PMID 29281947
- [Background] Maniam R, Tan MP, Chong MC. End of life care preference among hemodialysis population: Revisit Q methodology. Patient Educ Couns. 2022 Jun;105(6):1495-1502. doi: 10.1016/j.pec.2021.09.026. Epub 2021 Sep 29. PMID 34625322
- [Background] McLeod-Sordjan R. Death preparedness: a concept analysis. J Adv Nurs. 2014 May;70(5):1008-19. doi: 10.1111/jan.12252. Epub 2013 Sep 15. PMID 24102626
- [Background] Merces CAMF, Souto JDSS, Zaccaro KRL, de Souza JF, Primo CC, Brandao MAG. Death Anxiety: Concept Analysis and Clarification of Nursing Diagnosis. Int J Nurs Knowl. 2020 Jul;31(3):218-227. doi: 10.1111/2047-3095.12260. Epub 2019 Sep 20. PMID 31538748
- [Background] Miller-Lewis L, Tieman J, Rawlings D, Parker D, Sanderson C. Can Exposure to Online Conversations About Death and Dying Influence Death Competence? An Exploratory Study Within an Australian Massive Open Online Course. Omega (Westport). 2020 Jun;81(2):242-271. doi: 10.1177/0030222818765813. Epub 2018 Mar 26. PMID 29580148
- [Background] Nair D, Bonnet K, Wild MG, Umeukeje EM, Fissell RB, Faulkner ML, Bahri NS, Bruce MA, Schlundt DG, Wallston KA, Cavanaugh KL. Psychological Adaptation to Serious Illness: A Qualitative Study of Culturally Diverse Patients With Advanced Chronic Kidney Disease. J Pain Symptom Manage. 2021 Jan;61(1):32-41.e2. doi: 10.1016/j.jpainsymman.2020.07.014. Epub 2020 Jul 22. PMID 32711122
- [Background] Navise NH, Mokwatsi GG, Gafane-Matemane LF, Fabian J, Lammertyn L. Kidney dysfunction: prevalence and associated risk factors in a community-based study from the North West Province of South Africa. BMC Nephrol. 2023 Jan 30;24(1):23. doi: 10.1186/s12882-023-03068-7. PMID 36717778
- [Background] Nelson-Becker H, Victor C. Dying alone and lonely dying: Media discourse and pandemic conditions. J Aging Stud. 2020 Dec;55:100878. doi: 10.1016/j.jaging.2020.100878. Epub 2020 Sep 23. PMID 33272449
- [Background] O'Riordan J, Noble H, Kane PM, Smyth A. Advance care plan barriers in older patients with end-stage renal disease: a qualitative nephrologist interview study. BMJ Support Palliat Care. 2020 Dec;10(4):e39. doi: 10.1136/bmjspcare-2018-001759. Epub 2019 Jun 25. PMID 31239255
- [Background] Oskoui T, Pandya R, Weiner DE, Wong JB, Koch-Weser S, Ladin K. Advance Care Planning Among Older Adults With Advanced Non-Dialysis-Dependent CKD and Their Care Partners: Perceptions Versus Reality? Kidney Med. 2020 Jan 31;2(2):116-124. doi: 10.1016/j.xkme.2019.11.002. eCollection 2020 Mar-Apr. PMID 32734232
- [Background] Qiu Q, Zhang S, Lin X, Ban C, Yang H, Liu Z, Wang J, Wang T, Xiao S, Abdel-Khalek AM, Li X. Psychometric Properties of the Chinese Version of the Arabic Scale of Death Anxiety. Shanghai Arch Psychiatry. 2016 Jun 25;28(3):139-146. doi: 10.11919/j.issn.1002-0829.216033. PMID 28638183
- [Background] Raghavan D, Holley JL. Conservative Care of the Elderly CKD Patient: A Practical Guide. Adv Chronic Kidney Dis. 2016 Jan;23(1):51-6. doi: 10.1053/j.ackd.2015.08.003. PMID 26709063
- [Background] Rai NK, Wang Z, Drawz PE, Connett J, Murphy DP. CKD Progression Risk and Subsequent Cause of Death: A Population-Based Cohort Study. Kidney Med. 2023 Jan 21;5(4):100604. doi: 10.1016/j.xkme.2023.100604. eCollection 2023 Apr. PMID 36970224
- [Background] Richards CA, Liu CF, Hebert PL, Ersek M, Wachterman MW, Reinke LF, Taylor LL, O'Hare AM. Family Perceptions of Quality of End-of-Life Care for Veterans with Advanced CKD. Clin J Am Soc Nephrol. 2019 Sep 6;14(9):1324-1335. doi: 10.2215/CJN.01560219. Epub 2019 Aug 29. PMID 31466952
- [Background] Robbins RA. Death competency: a study of hospice volunteers. Death Stud. 1992 Nov-Dec;16(6):557-69. doi: 10.1080/07481189208252598. PMID 10122686
- [Background] Saeed F, Sardar MA, Davison SN, Murad H, Duberstein PR, Quill TE. Patients' perspectives on dialysis decision-making and end-of-life care . Clin Nephrol. 2019 May;91(5):294-300. doi: 10.5414/CN109608. PMID 30663974
- [Background] Sahan E, Eroglu MZ, Karatas MB, Mutluer B, Ugurpala C, Berkol TD. Death anxiety in patients with myocardial infarction or cancer. Egypt Heart J. 2018 Sep;70(3):143-147. doi: 10.1016/j.ehj.2018.04.003. Epub 2018 Apr 30. PMID 30190638
- [Background] Sellars M, Clayton JM, Detering KM, Tong A, Power D, Morton RL. Costs and outcomes of advance care planning and end-of-life care for older adults with end-stage kidney disease: A person-centred decision analysis. PLoS One. 2019 May 31;14(5):e0217787. doi: 10.1371/journal.pone.0217787. eCollection 2019. PMID 31150504
- [Background] Sellars M, Clayton JM, Morton RL, Luckett T, Silvester W, Spencer L, Pollock CA, Walker RG, Kerr PG, Tong A. An Interview Study of Patient and Caregiver Perspectives on Advance Care Planning in ESRD. Am J Kidney Dis. 2018 Feb;71(2):216-224. doi: 10.1053/j.ajkd.2017.07.021. Epub 2017 Nov 11. PMID 29132946
- [Background] Sharif Nia H, Pahlevan Sharif S, Koocher GP, Yaghoobzadeh A, Haghdoost AA, Mar Win MT, Soleimani MA. Psychometric Properties of the Death Anxiety Scale-Extended among Patients with End-Stage Renal Disease. Omega (Westport). 2020 Feb;80(3):380-396. doi: 10.1177/0030222817733220. Epub 2017 Oct 5. PMID 28982272
- [Background] Skulason B, Hauksdottir A, Ahcic K, Helgason AR. Death talk: gender differences in talking about one's own impending death. BMC Palliat Care. 2014 Mar 11;13(1):8. doi: 10.1186/1472-684X-13-8. PMID 24618410
- [Background] Soleimani MA, Bahrami N, Zarabadi-Pour S, Motalebi SA, Parker A, Chan YH. Predictors of death anxiety among patients with heart disease. Death Stud. 2020;44(3):160-167. doi: 10.1080/07481187.2018.1527416. Epub 2018 Nov 8. PMID 30407129
- [Background] Soleimani MA, Lehto RH, Negarandeh R, Bahrami N, Chan YH. Death Anxiety and Quality of Life in Iranian Caregivers of Patients With Cancer. Cancer Nurs. 2017 Jan/Feb;40(1):E1-E10. doi: 10.1097/NCC.0000000000000355. PMID 26925995
- [Background] Song MK, Ward SE, Fine JP, Hanson LC, Lin FC, Hladik GA, Hamilton JB, Bridgman JC. Advance care planning and end-of-life decision making in dialysis: a randomized controlled trial targeting patients and their surrogates. Am J Kidney Dis. 2015 Nov;66(5):813-22. doi: 10.1053/j.ajkd.2015.05.018. Epub 2015 Jun 30. PMID 26141307
- [Background] Templer DI. The construction and validation of a Death Anxiety Scale. J Gen Psychol. 1970 Apr;82(2d Half):165-77. doi: 10.1080/00221309.1970.9920634. No abstract available. PMID 4394812
- [Background] Uslu-Sahan F, Terzioglu F, Koc G. Hopelessness, Death Anxiety, and Social Support of Hospitalized Patients With Gynecologic Cancer and Their Caregivers. Cancer Nurs. 2019 Sep/Oct;42(5):373-380. doi: 10.1097/NCC.0000000000000622. PMID 29933308
- [Background] Van Scoy LJ, Green MJ, Reading JM, Scott AM, Chuang CH, Levi BH. Can Playing an End-of-Life Conversation Game Motivate People to Engage in Advance Care Planning? Am J Hosp Palliat Care. 2017 Sep;34(8):754-761. doi: 10.1177/1049909116656353. Epub 2016 Jul 12. PMID 27406696
- [Background] Van Scoy LJ, Levi BH, Witt P, Bramble C, Richardson C, Putzig I, Levi AR, Wasserman E, Chinchilli V, Tucci A, Green MJ. Association of Participation in an End-of-Life Conversation Game With Advance Care Planning Behavior and Perspectives Among African American Individuals. JAMA Netw Open. 2020 May 1;3(5):e204315. doi: 10.1001/jamanetworkopen.2020.4315. PMID 32383747
- [Background] Van Scoy LJ, Reading JM, Hopkins M, Smith B, Dillon J, Green MJ, Levi BH. Community Game Day: Using an End-of-Life Conversation Game to Encourage Advance Care Planning. J Pain Symptom Manage. 2017 Nov;54(5):680-691. doi: 10.1016/j.jpainsymman.2017.07.034. Epub 2017 Jul 23. PMID 28743662
- [Background] Van Scoy LJ, Reading JM, Scott AM, Chuang C, Levi BH, Green MJ. Exploring the Topics Discussed During a Conversation Card Game About Death and Dying: A Content Analysis. J Pain Symptom Manage. 2016 Nov;52(5):655-662. doi: 10.1016/j.jpainsymman.2016.03.021. Epub 2016 Sep 17. PMID 27650010
- [Background] Wasylynuk BA, Davison SN. An overview of advance care planning for patients with advanced chronic kidney disease: The basics. CANNT J. 2016 Jan-Mar;26(1):24-9. PMID 27215058
- [Background] Wen FH, Hsieh CH, Chou WC, Su PJ, Hou MM, Shen WC, Chen JS, Chang WC, Tang ST. Factors associated with cancer patients' distinct death-preparedness states. Psychooncology. 2023 Jul;32(7):1048-1056. doi: 10.1002/pon.6146. Epub 2023 Apr 27. PMID 37114337
- [Background] Yang CH, Wu CY, Low JTS, Chuang YS, Huang YW, Hwang SJ, Chen PJ. Exploring the Impact of Different Types of Do-Not-Resuscitate Consent on End-of-Life Treatments among Patients with Advanced Kidney Disease: An Observational Study. Int J Environ Res Public Health. 2021 Aug 2;18(15):8194. doi: 10.3390/ijerph18158194. PMID 34360487